CLINICAL TRIAL: NCT02877537
Title: Measurements of Change of Respiratory Admittance Induced by Salbutamol for Pediatric Asthma Diagnosis
Brief Title: Measurement of Respiratory Admittance for Pediatric Asthma Diagnosis
Acronym: SALBUTAMOL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2007-002822-31
Record Dates: First submitted 2016-08-19; First posted 2016-08-24 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Albuterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Asthma child (Experimental)
  Interventions: Drug: Salbutamol; Procedure: Forced oscillation technique; Procedure: Plethysmography
- Control adult (Experimental)
  Interventions: Drug: Salbutamol; Procedure: Forced oscillation technique; Procedure: Plethysmography
- Control child (Experimental)
  Interventions: Drug: Salbutamol; Procedure: Forced oscillation technique; Procedure: Plethysmography

INTERVENTIONS:
Drug: Salbutamol — bronchodilation obtained with 2 inhalations of salbutamol (100 µg per dose) with inhalation chamber
  Other Names: Ventoline
Procedure: Forced oscillation technique — before and after bronchodilation
Procedure: Plethysmography

SUMMARY:
The purpose is to characterize the change of respiratory admittance induced by salbutamol inhalation in children and young adults. A variation threshold will be fixed to distinguish asthmatic and healthy subjects.

This project could allow a better identification of asthmatic individuals needing a treatment, a reduction of morbidity of asthma, a reduction of unnecessary treatments administered in individuals with respiratory but not asthmatic symptoms, a better comprehension of bronchial hyperreactivity and its role in asthmatic disease.

ELIGIBILITY:
Inclusion Criteria:

Asthmatic children group:

* Several episodes of paroxysmal wheezes, spontaneous or after exercise, without bronchial-pulmonary infection
* Absence of bronchodilator taking during last 12 hours
* Absence of reported intolerance to adrenergic substances
* Parental authorization and consent of child to participate to the study

Control children group:

- Parental authorization and consent of child to participate to the study

Control adult group:

- Consent to participate to the study

Exclusion Criteria:

Control children and adult groups:

* At least 2 episodes of wheezes during breathing
* Several wheezes, abnormal breathlessness, cough during physical exercise
* Asthma diagnosed by family doctor
* Administration of drugs to treat asthma
* Eczema or food allergy at inclusion
* Episode of cough for longer than 6 weeks, without bronchial infection
* Bronchitis, throat infection, rhino-pharyngitis during last 15 days
* Paleness or cyanosis with loss of consciousness when the child was a baby or during an exercise

Ages: 3 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 177 (Actual)
Dates: Start 2008-10; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Ventilatory mechanical impedance | day 0
  Measured with Forced oscillation technique. 2 measures at basal status at 10 min interval for reproducibility and after 10 min broncodilation with salbutamol
Thoracic gas volume | day 0
  Measured with Plethysmography.

CONTACTS AND LOCATIONS:
Overall Officials: François MARCHAL, Principal Investigator — CHU de Nancy - Hôpital BRABOIS Enfants - Explorations fonctionnelles pédiatriques
Locations (1):
- CHU de Nancy - Hôpital BRABOIS Enfants - Explorations fonctionnelles pédiatriques, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No